CLINICAL TRIAL: NCT06172075
Title: Reducing Self-stigma and Increasing Treatment Seeking Intentions Among Youth With Depressive Symptoms: A Mixed-methods Study
Brief Title: Reducing Depression Self-stigma and Increasing Treatment Seeking Intentions Among Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Doron Amsalem, Assistant Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8366
Record Dates: First submitted 2023-11-18; First posted 2023-12-15 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Stigma, Social; Mental Health Disorder; Depression
MeSH Terms: conditions — Social Stigma; Mental Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Brief video intervention (Black Woman) (Experimental): A brief social contact-based video with a Black woman protagonist
  Interventions: Behavioral: Brief video intervention (Black Woman)
- Brief video intervention (Latinx Woman) (Experimental): A brief social contact-based video with a Latinx woman protagonist
  Interventions: Behavioral: Brief video intervention (Latinx Woman)
- Brief video intervention (White Woman) (Experimental): A brief social contact-based video with a White woman protagonist
  Interventions: Behavioral: Brief video intervention (White Woman)
- Vignette Control (Other): A brief vignette control condition
  Interventions: Behavioral: Vignette Control

INTERVENTIONS:
Behavioral: Brief video intervention (Black Woman) — A brief social contact-based video. The video presented a young Black woman in her early twenties, a professional actor, sharing her scripted personal story of struggles as a Black woman with depression and raising themes of recovery and hope.
  Arms: Brief video intervention (Black Woman)
Behavioral: Brief video intervention (Latinx Woman) — A brief social contact-based video. The video presented a young Latinx woman in her early twenties, a professional actor, sharing her scripted personal story of struggles as a Latinx woman with depression and raising themes of recovery and hope.
  Arms: Brief video intervention (Latinx Woman)
Behavioral: Brief video intervention (White Woman) — A brief social contact-based video. The video presented a young White woman in her early twenties, a professional actor, sharing her scripted personal story of struggles as a White woman with depression and raising themes of recovery and hope.
  Arms: Brief video intervention (White Woman)
Behavioral: Vignette Control — A brief vignette control condition with a script about a young woman who describes her struggles with depression and raises themes of recovery and hope.
  Arms: Vignette Control

SUMMARY:
Young people with depression, especially those of underserved minority groups, avoid treatment due to stigma and discrimination. Social contact is a form of interpersonal contact with members of the stigmatized group and the most effective type of intervention for improvement in stigma-related knowledge and attitudes.

In a prior study, the investigators developed short video interventions to reduce stigma and increase treatment seeking among people with depression. The videos vary by protagonist race/ethnicity (Latinx, non-Latinx Black, non-Latinx White) who share their experiences with depression, challenges, and recovery process. The investigators would like to test the efficacy of these videos using Prolific (a crowdsourcing platform). Specifically, the investigators are interested in conducting a randomized controlled trial (RCT) to test the efficacy of these videos as compared to a vignette control condition on reducing self-stigma and increasing help-seeking intentions and behavior at baseline, post, and 30 day follow-up among youth with depressive symptom scores on the PHQ-9≥ 5.

DETAILED DESCRIPTION:
In a randomized control trial (RCT) with pre-, post-intervention, and 30-day follow-up assessments, we aim to 1) test the efficacy of brief social video interventions, varying protagonist race/ethnicity, as compared to vignette control in reducing self-stigma and increasing treatment-seeking intentions and behavior among 1600 Prolific users ages 18-25 with depressive symptoms (PHQ-9≥ 5), and 2) explore whether matching to protagonist race/ethnicity increases intervention efficacy. We hypothesize that 1) Brief social contact-based video interventions will reduce self-stigma towards depression and increase treatment-seeking intentions and behavior compared to vignette control, and 2) The participants whose race/ethnicity match the protagonist will have greater changes in self-stigma and treatment-seeking than participants with unmatched protagonists, i.e., matching moderates the intervention's effects.

ELIGIBILITY:
Inclusion Criteria:

* Endorsing mild to severe depressive symptoms (Patient Health Questionnaire (PHQ-9) score of 5 or greater)
* Ages 18-25
* US Residents
* English speaking

Exclusion Criteria:

* Not endorsing mild to severe depressive symptoms
* Age less than 18 or greater than 25

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1520 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Depression Stigma | Baseline
  The Depression Stigma Scale (DSS) is a self-report scale comprised of two 9-item subscales measuring participants' personal beliefs about depression and participants' beliefs about others' attitudes (Griffiths et al., 2004). The current study will only utilize the personal beliefs subscale. Each item is rated on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). Scores range from 9 to 45. Higher scores indicate more stigma.
Depression Stigma | Post (immediately after the video or vignette control is shown)
  The Depression Stigma Scale (DSS) is a self-report scale comprised of two 9-item subscales measuring participants' personal beliefs about depression and participants' beliefs about others' attitudes (Griffiths et al., 2004). The current study will only utilize the personal beliefs subscale. Each item is rated on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). Scores range from 9 to 45. Higher scores indicate more stigma.
Depression Stigma | 30 day follow-up
  The Depression Stigma Scale (DSS) is a self-report scale comprised of two 9-item subscales measuring participants' personal beliefs about depression and participants' beliefs about others' attitudes (Griffiths et al., 2004). The current study will only utilize the personal beliefs subscale. Each item is rated on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). Scores range from 9 to 45. Higher scores indicate more stigma.
Attitude Towards Seeking Professional Psychological Help | Baseline
  Treatment seeking intentions will be measured using three items from the Attitudes Towards Seeking Professional Psychological Help Scale (ATSPPHS) Scale (Elhai et al., 2008). Items include: 'I might want to have psychological counselling in the future', 'I would want to get psychological help if I were worried or upset for a long period of time' and 'A person with an emotional problem is not likely to solve it alone; he or she is more likely to solve it with professional help'. Responses range from 1 (disagree) to 4 (agree). Total scores range from 3 to 12 with higher scores indicating higher treatment seeking intentions.
Attitude Towards Seeking Professional Psychological Help | Post (immediately after the video or vignette control is shown)
  Treatment seeking intentions will be measured using three items from the Attitudes Towards Seeking Professional Psychological Help Scale (ATSPPHS) Scale (Elhai et al., 2008). Items include: 'I might want to have psychological counselling in the future', 'I would want to get psychological help if I were worried or upset for a long period of time' and 'A person with an emotional problem is not likely to solve it alone; he or she is more likely to solve it with professional help'. Responses range from 1 (disagree) to 4 (agree). Total scores range from 3 to 12 with higher scores indicating higher treatment seeking intentions.
Attitude Towards Seeking Professional Psychological Help | 30 day follow-up
  Treatment seeking intentions will be measured using three items from the Attitudes Towards Seeking Professional Psychological Help Scale (ATSPPHS) Scale (Elhai et al., 2008). Items include: 'I might want to have psychological counselling in the future', 'I would want to get psychological help if I were worried or upset for a long period of time' and 'A person with an emotional problem is not likely to solve it alone; he or she is more likely to solve it with professional help'. Responses range from 1 (disagree) to 4 (agree). Total scores range from 3 to 12 with higher scores indicating higher treatment seeking intentions.
Treatment related stigma | Baseline
  Treatment-related stigma will be measured with the Self-Stigma of Seeking Help scale (SSOSH-3) (Brenner et al., 2021). Items include "I would feel inadequate if I went to a therapist for psychological help," "It would make me feel inferior to ask a therapist for help," and "If I went to a therapist, I would be less satisfied with myself." Response range from 1 (strongly disagree) to 5 (strongly agree). Total scores range from 3 to 15, with higher scores indicating greater stigma.
Treatment related stigma | Post (immediately after the video or vignette control is shown)
  Treatment-related stigma will be measured with the Self-Stigma of Seeking Help scale (SSOSH-3) (Brenner et al., 2021). Items include "I would feel inadequate if I went to a therapist for psychological help," "It would make me feel inferior to ask a therapist for help," and "If I went to a therapist, I would be less satisfied with myself." Response range from 1 (strongly disagree) to 5 (strongly agree). Total scores range from 3 to 15, with higher scores indicating greater stigma.
Treatment related stigma | 30 day follow-up
  Treatment-related stigma will be measured with the Self-Stigma of Seeking Help scale (SSOSH-3) (Brenner et al., 2021). Items include "I would feel inadequate if I went to a therapist for psychological help," "It would make me feel inferior to ask a therapist for help," and "If I went to a therapist, I would be less satisfied with myself." Response range from 1 (strongly disagree) to 5 (strongly agree). Total scores range from 3 to 15, with higher scores indicating greater stigma.
Actual help-seeking | 30 day follow-up
  One item will be utilized to measure actual help-seeking: Over the past 30 days, did you contact the mental health referrals we have provided or have sought out mental health treatment elsewhere?

SECONDARY OUTCOMES:
Emotional engagement | Post (immediately after the video or vignette control is shown)
  Emotional engagement will be measured using the Emotional Engagement Scale (de Vreede et al., 2019). The scale includes three items asking about emotional engagement (e.g., "I care about the contents of this video"), and response choices range from 1 (strongly disagree) to 4 (strongly agree). Total scores range from 3 to 12, with higher scores indicating greater emotional engagement.

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Griffiths KM, Christensen H, Jorm AF, Evans K, Groves C. Effect of web-based depression literacy and cognitive-behavioural therapy interventions on stigmatising attitudes to depression: randomised controlled trial. Br J Psychiatry. 2004 Oct;185:342-9. doi: 10.1192/bjp.185.4.342. PMID 15458995
- [Background] Elhai JD, Schweinle W, Anderson SM. Reliability and validity of the Attitudes Toward Seeking Professional Psychological Help Scale-Short Form. Psychiatry Res. 2008 Jun 30;159(3):320-9. doi: 10.1016/j.psychres.2007.04.020. Epub 2008 Apr 22. PMID 18433879
- [Background] Brenner RE, Colvin KF, Hammer JH, Vogel DL. Using Item Response Theory to Develop Revised (SSOSH-7) and Ultra-Brief (SSOSH-3) Self-Stigma of Seeking Help Scales. Assessment. 2021 Jul;28(5):1488-1499. doi: 10.1177/1073191120958496. Epub 2020 Sep 25. PMID 32975438
- [Background] de Vreede T, Andel SA, de Vreede GJ, Spector P, Singh V, Padmanabhan B. What is engagement and how do we measure it? Toward a domain independent definition and scale. Proceedings of the 52nd Hawaii International Conference on System Sciences. 2019, Hawaii. p. 749-758.